CLINICAL TRIAL: NCT00326651
Title: Home Usage of Conception Kit Instructions
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Conceivex (Industry)
Other Study IDs: Conception Kit
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Last update posted 2007-02-01 (Estimated); Status verified 2007-01

CONDITIONS: Healthy
Keywords: infertility; pregnancy; conception; conceive; conceiving; trying to conceive; get pregnant; conception kit; conception cap; fertility; Women who are actively trying to become pregnant
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

SUMMARY:
Patients will use the Conception Kit in their home and fill out a 22 question questionnaire in order to demonstrate their knowledge of the method of usage as described in the instructions and on the website: www.conceptionkit.com.

DETAILED DESCRIPTION:
Patients will be given a Conception Kit and take the Kit home and read the instructions and if needed consult the website. The patient will then complete a 22 question questionnaire in order to demonstrate their knowledge of the method of use.

All Components have 510K clearance. This study is a validation of the instructions for use (IFU) only.

OPK Class I Device 21CFR 862.1485, Conception Cap K993953, Pregnancy Test Kit K974059, Semen Collection Device K902936 (21CFR 884.5300),

Conception Kit has CE Marked by GMED. (Certificate 2037)

Conceivex is an ISO 13485: 2003 company

ELIGIBILITY:
Inclusion Criteria:

* Women who are actively trying to become pregnant

Exclusion Criteria:

* Women who are contraindicated for a pregnancy

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60
Dates: Start 2006-05; Study Completion 2007-05

CONTACTS AND LOCATIONS:
Overall Officials: Michael G La Vean, Study Director — Study Coordinator
Locations (2):
- United States (2):
  - Dr. Charles Barker, Belding, Michigan
  - Dr. Dorsey Ligon, Grand Rapids, Michigan

REFERENCES:
- [Background] Flierman PA, Hogerzeil HV, Hemrika DJ. A prospective, randomized, cross-over comparison of two methods of artificial insemination by donor on the incidence of conception: intracervical insemination by straw versus cervical cap. Hum Reprod. 1997 Sep;12(9):1945-8. doi: 10.1093/humrep/12.9.1945. PMID 9363712
- [Background] Coulson C, McLaughlin EA, Harris S, Ford WC, Hull MG. Randomized controlled trial of cervical cap with intracervical reservoir versus standard intracervical injection to inseminate cryopreserved donor semen. Hum Reprod. 1996 Jan;11(1):84-7. doi: 10.1093/oxfordjournals.humrep.a019044. PMID 8671164
- [Background] Subak LL, Adamson GD, Boltz NL. Therapeutic donor insemination: a prospective randomized trial of fresh versus frozen sperm. Am J Obstet Gynecol. 1992 Jun;166(6 Pt 1):1597-604; discussion 1604-6. doi: 10.1016/0002-9378(92)91548-o. PMID 1615966
- [Background] Williams DB, Moley KH, Cholewa C, Odem RR, Willand J, Gast MJ. Does intrauterine insemination offer an advantage to cervical cap insemination in a donor insemination program? Fertil Steril. 1995 Feb;63(2):295-8. doi: 10.1016/s0015-0282(16)57358-0. PMID 7843434
- [Background] Corrigan E, McLaughlin EA, Coulson C, Ford WC, Hull MG. The effect of halving the standard dose of cryopreserved semen for donor insemination: a controlled study of conception rates. Hum Reprod. 1994 Feb;9(2):330-3. doi: 10.1093/oxfordjournals.humrep.a138502. PMID 8027291
- [Background] Perino A, Cimino C, Catinella E, Barba G, Cittadini E. In vitro sperm capacitation and intrauterine insemination (IVC-Insem): a simple technique for the treatment of refractory infertility unrelated to female organic pelvic disease. Clinical results and immunological effects: a preliminary report. Acta Eur Fertil. 1986 Sep-Oct;17(5):325-31. PMID 3577597
- [Background] Corson SL, Batzer FR, Otis C, Fee D. The cervical cap for home artificial insemination. J Reprod Med. 1986 May;31(5):349-52. PMID 3746786
- [Background] Noci I, Chelo E, Scarselli G, Messori A. Cervical cap homologous artificial insemination (AIH): the University of Florence experience. Acta Eur Fertil. 1986 Mar-Apr;17(2):133-7. PMID 3739559
- [Background] Bergquist CA, Rock JA, Miller J, Guzick DS, Wentz AC, Jones GS. Artificial insemination with fresh donor semen using the cervical cap technique: a review of 278 cases. Obstet Gynecol. 1982 Aug;60(2):195-9. PMID 7155481
- [Background] Carruthers GB. Present-day management of male infertility. IPPF Med Bull. 1982 Jun;16(3):1-2. PMID 12338236
- [Background] Coucke W, Steeno O. Pregnancy rate after homologous insemination. Arch Androl. 1979;2(1):73-6. doi: 10.3109/01485017908987295. PMID 443924
- [Background] Segal S, Sherer M. The use of donor mucus and insemination for cervical factor. Int J Fertil. 1979;24(4):291-2. PMID 45104
- [Background] Jondet D, Millet D, Netter A. [Adaptation of a cervical cap for human artificial insemination]. J Gynecol Obstet Biol Reprod (Paris). 1975 Jan-Feb;4(1):141-4. French. PMID 1230473
- [Background] Meyer WR, Smith PM, Clark MR, Cusmano LL, Fritz MA. Therapeutic cup insemination with cryopreserved donor sperm: prognostic value of cervical mucus score at insemination and the number of motile sperm in mucus at 24 hours. Fertil Steril. 1996 Sep;66(3):435-9. doi: 10.1016/s0015-0282(16)58515-x. PMID 8751744
- [Background] Drobnis EZ, Clisham PR, Brazil CK, Wisner LW, Zhong CQ, Overstreet JW. Detection of altered acrosomal physiology of cryopreserved human spermatozoa after sperm residence in the female reproductive tract. J Reprod Fertil. 1993 Sep;99(1):159-65. doi: 10.1530/jrf.0.0990159. PMID 8283434
- [Background] Depypere HT, Gordts S, Campo R, Comhaire F. Methods to increase the success rate of artificial insemination with donor semen. Hum Reprod. 1994 Apr;9(4):661-3. doi: 10.1093/oxfordjournals.humrep.a138567. PMID 8046019
- [Background] Diamond MP, Christianson C, Daniell JF, Wentz AC. Pregnancy following use of the cervical cup for home artificial insemination utilizing homologous semen. Fertil Steril. 1983 Apr;39(4):480-4. doi: 10.1016/s0015-0282(16)46936-0. PMID 6832404
- [Background] Scott JZ, Nakamura RM, Mutch J, Davajan V. The cervical factor in infertility: diagnosis and treatment. Fertil Steril. 1977 Dec;28(12):1289-94. doi: 10.1016/s0015-0282(16)42971-7. PMID 590536
- [Background] Hanson FW, Overstreet JW. The interaction of human spermatozoa with cervical mucus in vivo. Am J Obstet Gynecol. 1981 May 15;140(2):173-8. doi: 10.1016/0002-9378(81)90105-8. PMID 7234912
- [Background] O'Brien P, Vandekerckhove P. Intra-uterine versus cervical insemination of donor sperm for subfertility. Cochrane Database Syst Rev. 2000;(2):CD000317. doi: 10.1002/14651858.CD000317. PMID 10796709
- [Result] Mahony MC. Evaluation of the effect of a cervical cap device on sperm functional characteristics in vitro. Andrologia. 2001 Jul;33(4):207-13. doi: 10.1046/j.1439-0272.2001.00426.x. PMID 11472332
- [Result] Adamson GD, Subak LL, Boltz NL, McNulty MA. Failure of intrauterine insemination in a refractory infertility population. Fertil Steril. 1991 Aug;56(2):361-3. doi: 10.1016/s0015-0282(16)54502-6. PMID 2070868